CLINICAL TRIAL: NCT06274242
Title: Mixed Natural Prebiotic-Fibers Impact on Stool Frequency and Fecal Microbiota in Constipated Thai Adults: A Randomized Clinical Trial.
Brief Title: Mixed Natural Prebiotic-Fibers Impact on Stool Frequency and Fecal Microbiota in Constipated Thai Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirirat Luk-In, Assistant professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-CIRB 2022/300.0711
Record Dates: First submitted 2024-02-13; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic arm (Experimental)
  Interventions: Dietary Supplement: Haruna
- Placebo arm (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Haruna — Mixed Natural Prebiotic-Fibers (Ginkgo nut, Spinach, Corn, Brown rice)
  Arms: Prebiotic arm
Dietary Supplement: Placebo Powder — Isolate Soy Protein and Isomalt
  Arms: Placebo arm

SUMMARY:
Mixed Natural Prebiotic-Fibers Impact on Stool Frequency and Fecal Microbiota in Constipated Thai Adults: A Randomized Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with a Body mass index (BMI) of 16.00 to 29.99 kg/m2
* Self-reported constipation according to the Rome IV criteria

Exclusion Criteria:

* Pregnancy
* Crohn's disease or any other inflammatory bowel disease
* Pelvic floor dyssynergia
* Have congenital diseases such as liver disease, diabetes, and thyroid dysfunction. hypercalcemia neurological disease
* Drink alcohol or smoke regularly.
* During the past 1 month or while in the project, have received antibiotics, steroids, NSAIDs, blood pressure-lowering drugs, antidepressants, anticonvulsants, or Parkinson's disease medications
* History of food allergy to Haruna's ingredients
* There has been a change in body weight (increase or decrease of 5 kilograms over a period of 6 months).
* During the past 2 weeks or while in the project, have received probiotics or other prebiotics

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
Change in Stool Frequency | 12 weeks
  Stool frequency during the intervention period was determined by modified Constipation scoring system using questionnaire with the following variables: frequency of bowel movements; painful evacuation effort; feeling of incomplete evacuation; abdominal pain; minutes in lavatory per attempt; type of assistance; unsuccessful attempts for evacuation. This consists of six items that are scored using a five-point Likert scale that ranges from 0 (none of the time) to 4 (all of the time) and one item that is rated on a 0-2 scale. A total score can range from 0 (normal) to 26 (severe constipation).
Change in Fecal Microbiota | 12 weeks
  Change in Bifidobacterium relative abundance with 2log ratio of relative abundance, during the intervention period, compared between prebiotic arm and placebo arm. Subjects with an increase in Bifidobacterium relative abundance were considered to have a good response.

SECONDARY OUTCOMES:
Change in Stool consistency | 12 weeks
  Stool consistency during the intervention period was determined by Bristol stool scale score using questionnaire with the following scale score: 1, separate hard lumps, like nuts; 2, sausage-shaped but lumpy; 3, like a sausage but with cracks on its surface; 4, like a sausage or snake, smooth and soft; 5, soft blobs with clear-cut edges; 6, fluffy pieces with ragged edges, a mushy stool; 7, watery, no solid pieces. 1-2 scale indicate constipation. 3-4 scale are ideal stools as they are easier to pass. 5-7 scale may indicate diarrhea and urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Luk-in, phD, Principal Investigator — Department of Clinical Microbiology and Applied Technology, Faculty of Medical Technology, Mahidol University
Locations (1):
- Mahidol University, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Yes
After the publication of this research project.
Supporting Information: Study Protocol
Time Frame: After the publication of this research project.